CLINICAL TRIAL: NCT00003351
Title: Randomized Phase II Trial of Irinotecan (CPT-11) In Patients With Refractory Metastatic Breast Cancer
Brief Title: Irinotecan in Treating Patients With Refractory Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-963255; CDR0000066332 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-03-01 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: irinotecan (Experimental): Patients receive irinotecan intravenously over 90 minutes every week for 4 weeks followed by a 2 week rest period. Treatment is repeated every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed before and during treatment. Patients are followed every 3 months for 2 years, then annually for 1 year.
  Interventions: Drug: irinotecan hydrochloride
- Arm II: irinotecan (Experimental): Patients receive irinotecan intravenously over 90 minutes every 3 weeks for 6 weeks. Treatment is repeated every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed before and during treatment. Patients are followed every 3 months for 2 years, then annually for 1 year.
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to compare the effectiveness of two regimens of irinotecan in treating patients who have refractory metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity and toxicity of two different schedules of irinotecan in the treatment of patients with refractory metastatic breast cancer who have received 1 or 2 previous chemotherapy regimens (up to one prior therapy for metastatic disease and one for adjuvant therapy). II. Compare the time to progression, survival, and quality of life of these patients on these 2 different schedules of irinotecan.

OUTLINE: This is a randomized study. Patients are stratified according to dominant disease (visceral vs nonvisceral), performance status (0-1 vs 2), and prior chemotherapy in metastatic setting (yes vs no). Patients assigned to arm I receive irinotecan intravenously over 90 minutes every week for 4 weeks followed by a 2 week rest period. Treatment is repeated every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients assigned to arm II receive irinotecan intravenously over 90 minutes every 3 weeks for 6 weeks. Treatment is repeated every 6 weeks in the absence of disease progression or unacceptable toxicity. Quality of life is assessed before and during treatment. Patients are followed every 3 months for 2 years, then annually for 1 year.

PROJECTED ACCRUAL: A total of 42-100 patients (21-50 patients per arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the breast with progressing locoregional or metastatic disease Measurable or evaluable indicator lesion No uncontrolled CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 0.3 mg/dL above upper limit of normal (ULN) AST no greater than 3 times ULN Renal: Creatinine no greater than 1.0 mg/dL above ULN Cardiovascular: No New York Heart Association class III or IV heart disease Other: No uncontrolled infection No chronic debilitating disease Not pregnant or lactating Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since chemotherapy No more than 2 prior chemotherapy regimens for metastatic disease No more than 1 prior chemotherapy regimen in the adjuvant setting At least 1 prior regimen containing taxane or doxorubicin for metastatic disease or in the adjuvant setting Endocrine therapy: Not specified Radiotherapy: No radiotherapy to greater than 25% of bone marrow No prior treatment with strontium 89 Surgery: At least 4 weeks since major surgery Other: No concurrent metoclopramide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 1998-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Time to progression | Up to 3 years

SECONDARY OUTCOMES:
Survival | Up to 3 years
Quality of life | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (22):
- United States (21):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Perez EA, Hillman DW, Milliard JA, et al.: Randomized phase II study of 2 schedules of irinotecan (CPT-11) for patients (pts) with refractory metastatic breast cancer (MBC): an NCCTG Cooperative Group study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-206, 2002.